CLINICAL TRIAL: NCT00805974
Title: Study of the Relationship Between Sleep Quality and Daytime-Nighttime Variations of Blood Pressure and Plasma Glucose Type I
Acronym: DIAPASOM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties for including diabetic patients
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Pr Mallion Jean-Michel (Unknown); Pr BAGUET Jean-Philippe (Unknown); Pr BENHAMOU Pierre-Yves (Unknown); Pr LEVY Patrick (Unknown); Dr MOURET Sandrine (Unknown); Dr ORMEZZANO Olivier (Unknown); Pr PEPIN Jean-Louis (Unknown); Dr TAMISIER Renaud (Unknown)
Responsible Party: Pr MALLION Jean-Michel, Professor, PhD,, University Hospital, Grenoble
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0513; 2005/0479
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Type 1 Diabetes
Keywords: diapasom; sleep quality; type I diabete; blood pressure; plasma glucose; daytime and nighttime variations
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Sleep Initiation and Maintenance Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Biological examinations (blood and urinary).

SUMMARY:
The primary objectives are to compare the mean levels of the sleep quality parameters of subjects : with a nocturnal fall of the SBP (Systolic blood pressure), DBP (diastolic blood pressure) and MAP (mean arterial pressure) over of egal to 10% (dipping subjects) and of subjects with a nocturnal fall of SBP, DBP and MAP inferior to 10% (non dipper subjects).

The secondary objectives are :

Establish correlations between:

* The quality of sleep parameters
* The parameters of BP variations between the diurnal and nocturnal periods and the awake periods of sleep defined in reference to polysomnography.
* The glycemia levels on 24h with a glycemic holter. The parameters of the sympathic system activation evaluated in reference to the measure of the baroreflex sensibility during the awake period.

DETAILED DESCRIPTION:
It is a prospective monocentric study after a preliminary period of depistage of the sleep abnormalities by oximetry at home. The patient would be hospitalized for two consecutive days (J0, J1). And the following evaluations will be done:

* Nocturnal oxymetric + Epworth questionnaire + clinical questionnaire to detect sleep perturbations at home.
* Blood pressure + heart rate measure
* Ambulatory blood pressure monitoring on 24 hours
* Polysomnographic measurements during the J0-J1 night spend at the hospital.
* Questionnaire of sleep quality and of quality of life.
* Glycemic measurements on 24h (J0-J1).
* Measure of the baroreflex sensibility during the awake period at J1.
* Electrocardiogram
* Biological examinations (blood and urinary).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 60 years of age
* Who have given their written consent to participate in this study
* Who are affiliated to the French social security system
* Are able to travel to Grenoble University Hospital
* Type I diabetes in reference to the 1997 criteria (American Diabetes Association) without any recent cetoacidosis or severe hypoglycaemia during the previous month and with a HbA1c < 10% during the previous month.
* Normal blood pressure or essential hypertension light or moderate (SBP) at rest in the sitting position >= 140 mmHg and < 180 mmHg and/or PAD >= 90 mmHg et < 110 mmHg), with or without treatment.

Exclusion Criteria:

* Non stabilised diabetes with at least one episode of acidoketosis decompensation or hypoglycemic coma during the previous month.
* Diabetic nephropathy patent stage 4 with a creatinine > 150 mol / L and / or creatinine clearance <50 ml / min
* Diabetic nephropathy in evolution
* Severe hypertension (SBP at rest in the sitting position >= 180 mmHg and/or DBP >= 110 mmHg)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Polysomnographic measurements during the D0-D1 night spend at the hospital | inclusion visit
Ambulatory blood pressure monitoring on 24 hours | inclusion visit

SECONDARY OUTCOMES:
Glycemic measurements on 24h (D0-D1). | inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: MALLION Jean-Michel, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France

REFERENCES:
- [Derived] Borel AL, Benhamou PY, Baguet JP, Halimi S, Levy P, Mallion JM, Pepin JL. High prevalence of obstructive sleep apnoea syndrome in a Type 1 diabetic adult population: a pilot study. Diabet Med. 2010 Nov;27(11):1328-9. doi: 10.1111/j.1464-5491.2010.03096.x. No abstract available. PMID 20950392